CLINICAL TRIAL: NCT00676728
Title: A Phase 1 Study of the Histone-deacetylase Inhibitor JNJ-26481585 in Subjects With Advanced or Refractory Leukemia or Myelodysplastic Syndrome
Brief Title: A Study of the Histone-deacetylase Inhibitor JNJ-26481585 in Patients With Advanced or Refractory Leukemia or Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013960; 26481585CAN1003 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Advanced or Refractory Leukemia; Myelodysplastic Syndromes
Keywords: Advanced or Refractory Leukemia; Myelodysplastic Syndromes; JNJ 26481585; Histone-Deacetylase Inhibitor; Advanced Leukemia; Refractory Leukemia
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — quisinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JNJ-26481585 (Experimental)
  Interventions: Drug: JNJ-26481585

INTERVENTIONS:
Drug: JNJ-26481585 — In Part 1, Initial dose of JNJ-26481585 4 mg oral capsule is administered once daily on each day of a 21-day cycle. Dose will be escalated or de-escalated until Maximum tolerated dose (MTD) of JNJ-26481585 is determined in Part 1. MTD of JNJ-26481585 will be the initial dose in Part 2.

SUMMARY:
The purpose of this study is to explore the safety, pharmacokinetic (what the body does to the medication), pharmacodynamic (what the medication does to the body), and activity of JNJ-26481585 in patients with advanced or refractory leukemia and myelodysplastic syndrome (MDS).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), Phase 1 dose escalation, 2-part study (Part I and Part II). In Part I of the study, the Maximum Tolerated Dose (MTD) defined as the highest dose with an observed incidence of dose limiting toxicity (DLT) in no more than 1 in 6 patients, will be determined using rapid escalation (Stage 1) followed by conventional escalation (Stage 2). In Stage 1, at least 2 patients will be enrolled at each dose level; dose increments of 100% will be applied. In Stage 2, at least 3 patients will be enrolled at each dose level and dose increments of 20-50% will be implemented. Decisions on dose escalation or de-escalation, changes in the timing of pharmacokinetic/pharmacodynamic sampling, and the exploration of an alternative schedule were to be made by the Study Evaluation Team (SET), which consisted of all principal investigators, the medical monitor, and 1 of the sponsor's clinical pharmacologists. Part II of the study will be the expansion phase, which will begin after the MTD had been determined in Part I and an additional cohort of patients with MDS will be enrolled to further explore the safety and activity of JNJ 26481585 in patients with MDS. The starting dose for patients enrolled in Part II of the study was to be the MTD established in Part I. Depending on the outcome, the SET may decide to continue at the MTD dose, or dose-de-escalate to the next lower level (25 50% decrement from MTD). The cohort for MDS will be expanded to consist of 16 evaluable patients. Safety will be evaluated throughout the study and will include evaluations of adverse events clinical laboratory tests, electrocardiogram (ECG), vital signs, 24 hours Holter ECG, physical examination, Eastern Cooperative Oncology Group performance status and Multiple Gated Acquisition scan or echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced or refractory acute myeloid leukemia, acute lymphocytic leukemia, chronic myeloid leukemia in blast phase, refractory chronic lymphocytic leukemia, myelodysplastic syndrome, or chronic myelomonocytic leukemia
* For Part II, patients with myelodysplastic syndrome
* Eastern Cooperative Oncology Group Performance Status Score 0, 1 or 2
* Left Ventricular Ejection Fraction greater than or equal to 50%
* Negative hepatitis B, C and human immunodeficiency virus (HIV) test within last 3 months
* Adequate liver and kidney function

Exclusion Criteria:

* Known or suspected involvement of the central nervous system
* Chemotherapy (nitrosoureas and mitomycin C within 6 weeks), radiotherapy, immunotherapy or treatment with investigative agent within 3 weeks before study drug administration (except hydroxyurea which should be stopped at least 24 hours prior to first dose)
* Unstable angina or myocardial infarction within the preceding 12 months; congestive heart failure
* Poorly controlled hypertension or diabetes, ongoing active infection and psychiatric illness
* Receiving medications known to have a risk of causing QTc prolongation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | Upto 14 days after last dose administration of study medication
Number of patients with dose limiting toxicity [DLT] | From the date of dosing upto 3 months after the date the last patient enrolled in Part I of the study, received the first dose of study medication
  Only toxicities that occur during Treatment Cycle 1 will be used for the purposes of defining DLT.
Maximum tolerated dose (MTD) of JNJ 26481585 | From the date of dosing upto 3 months after the date the last patient enrolled in Part I of the study, received the first dose of study medication
  The MTD is defined as the highest dose with an observed incidence of DLT in no more than 1 in 6 patients.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of JNJ 26481585 | Days 1, 2, 8, 15 and 21 of Cycle 1
Time to reach maximum plasma concentration (tmax) of JNJ-26481585 | Days 1, 2, 8, 15 and 21 of Cycle 1
Area under the plasma concentration-time curve from time 0 to 24 hours (AUC0-24) | Days 1, 2, 8, 15 and 21 of Cycle 1
Elimination half-life (t1/2) of JNJ-26481585 | Days 1, 2, 8, 15 and 21 of Cycle 1
Cumulative amount of drug excreted in urine over 24 hours (Ae24) | Days 1 and 21 of Cycle 1
Renal clearance (CLR) of JNJ 26395018 | Days 1 and 21 of Cycle 1
Concentration of biomarker histone acetylation | Days 1 and 21 of Cycle 1; Day 21 of Cycles 2 to 20
Concentration of biomarker interleukin-6 (IL-6) | Days 1 and 21 of Cycle 1; Day 21 of Cycles 2 to 20
Concentration of biomarker heat shock protein 90 (Hsp90) | Days 1 and 21 of Cycle 1; Day 21 of Cycles 2 to 20
Complete Blood Count (CBC) | Pre-treatment (within 4 weeks prior to first dose of JNJ-26481585); Days 1, 3, 8, 15 and 21 of Cycle 1; Days 8, 15 and 21 of Cycle 2; Day 21 of Cycle 3 to 20; follow up (within 14 days after last dose of JNJ-26481585)
  Anticancer activity of JNJ-26481585 explored by assessment of response parameters such as CBC.
Assessment of Transfusion Record | From Day 1 of Cycle 1 upto 14 days after last dose
  Assessment of Transfusion Record is the parameter for assessment of response.
Radiological Tumor Mass assessment | Pre-treatment, Day 21 of Cycle 2 to 20 and follow up
  Radiological Tumor Mass assessment is the parameter for assessment of response.
Bone marrow aspirate/biopsy assessment | Pre-treatment, Day 21 of Cycles 1 to 20
  Bone marrow aspirate/biopsy assessment is the parameter for assessment of response.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (2):
- United States (2):
  - Baltimore, Maryland
  - Houston, Texas

REFERENCES:
- See also: A Phase 1 Study of the Histone-Deacetylase Inhibitor JNJ-26481585 in Subjects with Advanced or Refractory Leukemia or Myelodysplastic Syndrome — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=766&filename=CR013960_CSR.pdf